CLINICAL TRIAL: NCT03074149
Title: Investigating Idiopathic Pulmonary Fibrosis in Greece
Acronym: INDULGEIPF
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199.252
Record Dates: First submitted 2017-01-04; First posted 2017-03-08 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic Pulmonary Fibrosis (IPF) patients with less than 6 months diagnosis
- Idiopathic Pulmonary Fibrosis (IPF) patients with equal or more than 6 months diagnosis

SUMMARY:
To gain further insight on the characteristics, management, disease progression and the outcomes of patients with IPF, as diagnosed and treated under real-world, clinical practice conditions in Greece. More specifically, this registry will be used to: Provide a comprehensive clinical picture of IPF, Track access to health care and cost of caring for IPF patients over time, Examine the implementation of treatment guidelines used on patients diagnosed with IPF, according to the existing diagnosis guidelines, Characterization of patients on different treatments. To provide information regarding survival and mortality causes, IPF exacerbations as well as IPF patient co-morbidities including myocardial infarction, CNS infarction, other arterial thromboembolic events, deep vein thrombosis, hemorrhage, gastrointestinal perforation and pulmonary hypertension. Data regarding IPF patient hospitalization will be collected and evaluated with regards to potential respiratory causes, and there will be documentation of treatment patterns and economic aspects. Patients will be followed up for 2 years and information regarding IPF treatment changes since the last visit will be collected.

DETAILED DESCRIPTION:
Purpose: To gain further knowledge on the characteristics, management, progression and outcomes of patients with IPF as treated under real-world, clinical practice conditions in Greece

Study Design:

National, multi-center, observational disease registry based on new data from a significant sample size of IPF patients in Greece. Patients will be followed up for 2 years and information will be collected during this time period. This is a non-interventional study and primary data collected during study visits will be used

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed (less than 6 months) or patients previously diagnosed with IPF (more than 6 months from baseline visit), based upon the consensus statement jointly issued by ATS/ERS/JRS/ALAT in 2011 (see Annexes 6 and 7 for HRCT and histological criteria in Annex 6)

  * Exclusion of other known causes of ILD (e.g., domestic and occupational environmental exposures, connective tissue disease, and drug toxicity)
  * Assessment of IPF based on HRCT or combinations of HRCT and surgical lung biopsy, if available
* Age =40 years old at the time of inclusion
* Written informed consent for participation in the registry
* Patients that can be followed up further, during the scheduled study period

Exclusion criteria:

* Expected lung transplantation within the following 6 months
* Participation in clinical trials

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible for participation in the study patients must fulfill ALL the inclusion criteria and NONE of the exclusion criteria that are listed below and must be consecutively enrolled:
  * Newly diagnosed (less than 6 months) or patients previously diagnosed with IPF (more than 6 months from baseline visit), based upon the consensus statement jointly issued by ATS/ERS/JRS/ALAT in 2011
    * Exclusion of other known causes of ILD (e.g., domestic and occupational environmental exposures, connective tissue disease, and drug toxicity)
    * Assessment of IPF based on HRCT or combinations of HRCT and surgical lung biopsy, if available
  * Age ≥40 years old at the time of inclusion
  * Written informed consent for participation in the registry
  * Patients that can be followed up further, during the scheduled study period
  None of the following Exclusion Criteria should be fulfilled:
  * Expected lung transplantation within the following 6 months
  * Participation in clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Greece (7):
  - Gen. Hosp. of Chest Diseases "Sotiria", Univ. Resp. Med., Athens
  - Sotiria Hospital Athens, 7th Pulmonary Clinic, Athens
  - University General Hospital Attikon, Athens
  - University Hospital of Heraklion, University Pulmonology Cl, Heraklion
  - General University Hospital of Larissa, Larissa
  - A Pulmonology Clinic "G.Papanikolaou" Hospital Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data- 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a national, multi -center, observational disease and outcomes registry study based on new data from a significant sample size of Greek idiopathic pulmonary fibrosis (IPF) patients.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- IPF Patients With Less Than 6 Months Diagnosis: Patients in Greece diagnosed less than 6 months (newly diagnosed) with Idiopathic Pulmonary Fibrosis (IPF) from the study baseline visit.
- IPF Patients With Equal or More Than 6 Months Diagnosis: Patients in Greece diagnosed since 6 or more months with Idiopathic Pulmonary Fibrosis (IPF) from the study baseline visit.
Period: Overall Study
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Started | 96 | 205
Completed | 64 | 125
Not Completed | 32 | 80
Not completed — Reason unknown | 22 | 35
Not completed — Death | 10 | 45

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) comprised of all subjects enrolled in the study with at least one measurement of any of the primary endpoints during the study. This population was used to run any statistics of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis | Total
Number analyzed (Participants) | 96 | 205 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.4 (7.27) | 70.8 (7.87) | 71.6 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 37 | 55
  Male | 78 | 168 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 96 | 205 | 301
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Category of Non-pharmacological Treatment for Idiopathic Pulmonary Fibrosis (IPF) by Study Visit
Description: Number in each category of non-pharmacological treatment (e.g. start of Long-term oxygen therapy (LTOT), new listing for lung transplantation, physiotherapy) for Idiopathic Pulmonary Fibrosis (IPF) by study visit is reported.
  The categories of non-pharmacological treatment for Idiopathic Pulmonary Fibrosis (IPF) are the following:
  * No
  * Yes
  * Unknown
  * Missing
Time Frame: At baseline visit and at 3 months, at 6 months, at 12 months, at 18 months and at 24 months after the baseline visit.
Population: Full Analysis Set (FAS) comprised all subjects enrolled in the study with at least one measurement of any of the primary endpoints during the study. This population was used to run any statistics of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Number analyzed (Participants) | 96 | 205
Participants
  Baseline: No | 83 | 162
  Baseline: Yes | 13 | 43
  Baseline: Unknown | 0 | 0
  Baseline: Missing | 0 | 0
  3 months: No | 70 | 137
  3 months: Yes | 13 | 37
  3 months: Unknown | 3 | 1
  3 months: Missing | 10 | 30
  6 months: No | 67 | 127
  6 months: Yes | 11 | 35
  6 months: Unknown | 2 | 7
  6 months: Missing | 16 | 36
  12 months: No | 66 | 116
  12 months: Yes | 10 | 38
  12 months: Unknown | 0 | 7
  12 months: Missing | 20 | 44
  18 months: No | 61 | 109
  18 months: Yes | 10 | 29
  18 months: Unknown | 2 | 2
  18 months: Missing | 23 | 65
  24 months: No | 55 | 96
  24 months: Yes | 9 | 27
  24 months: Unknown | 0 | 2
  24 months: Missing | 32 | 80

2. Primary Outcome: Number of Patients in Each Category of Physician's Clinical Assessment of the Probable Course of Idiopathic Pulmonary Fibrosis (IPF) by Study Visit
Description: Number of patients in each category of physician's clinical assessment of the probable course of IPF by study visit is reported. Physician's clinical rating of the probable course of IPF (stable, slow or rapid progression) was based on available Forced vital capacity (FVC) results, diffusion capacity for carbon monoxide (DLCO) results, physical examination, hospitalizations/events between the visits. The categories of physician's clinical assessment are the following:
  * Stable disease
  * Slow progression
  * Rapid progression
  * No judgement possible
  * Missing
Time Frame: At baseline (up to 12 months prior to baseline visit) and at 3 months, at 6 months, at 12 months, at 18 months and at 24 months after the baseline visit.
Population: Full Analysis Set (FAS) comprised all subjects enrolled in the study with at least one measurement of any of the primary endpoints during the study. This population was used to run any statistics of the study. Only participants with non-missing results are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Number analyzed (Participants) | 96 | 205
Participants
  Baseline (up to 12 months prior to baseline visit): Stable disease | 79 | 158
  Baseline (up to 12 months prior to baseline visit): Slow progression | 13 | 41
  Baseline (up to 12 months prior to baseline visit): Rapid progression | 2 | 3
  Baseline (up to 12 months prior to baseline visit): No judgement possible | 2 | 3
  Baseline (up to 12 months prior to baseline visit): Missing | 0 | 0
  3 months (since last visit): Stable disease | 75 | 156
  3 months (since last visit): Slow progression | 7 | 16
  3 months (since last visit): Rapid progression | 3 | 3
  3 months (since last visit): No judgement possible | 1 | 0
  3 months (since last visit): Missing | 10 | 30
  6 months (since last visit): Stable disease | 71 | 140
  6 months (since last visit): Slow progression | 4 | 23
  6 months (since last visit): Rapid progression | 5 | 6
  6 months (since last visit): No judgement possible | 0 | 0
  6 months (since last visit): Missing | 16 | 36
  12 months (since last visit): Stable disease | 64 | 134
  12 months (since last visit): Slow progression | 10 | 22
  12 months (since last visit): Rapid progression | 2 | 3
  12 months (since last visit): No judgement possible | 0 | 2
  12 months (since last visit): Missing | 20 | 44
  18 months (since last visit): Stable disease | 63 | 113
  18 months (since last visit): Slow progression | 6 | 21
  18 months (since last visit): Rapid progression | 4 | 5
  18 months (since last visit): No judgement possible | 0 | 0
  18 months (since last visit): Missing | 23 | 66
  24 months (since last visit): Stable disease | 50 | 100
  24 months (since last visit): Slow progression | 10 | 21
  24 months (since last visit): Rapid progression | 4 | 4
  24 months (since last visit): No judgement possible | 0 | 0
  24 months (since last visit): Missing | 32 | 80

3. Primary Outcome: Number of Physician Contacts Per Patient by Study Visit
Description: Number of physician contacts per patient is reported. For the baseline visit mean and standard deviation of physician contacts with the patient up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months mean and standard deviation of physician contacts with the patient since the last study visit is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: physician contacts per patient
Groups:
- Idiopathic Pulmonary Fibrosis Diagnosed Patients: This arm includes all Idiopathic Pulmonary Fibrosis (IPF) diagnosed patients in Greece who participated in this study.
Arm/Group | Idiopathic Pulmonary Fibrosis Diagnosed Patients
Number analyzed (Participants) | 301
physician contacts per patient
  Baseline (up to 12 months prior to baseline visit) | 3.651 (2.506)
  3 months (since last visit): number analyzed (Participants) | 261
  3 months (since last visit) | 0.801 (1.033)
  6 months (since last visit): number analyzed (Participants) | 247
  6 months (since last visit) | 0.676 (0.832)
  12 months (since last visit): number analyzed (Participants) | 237
  12 months (since last visit) | 1.105 (1.406)
  18 months (since last visit): number analyzed (Participants) | 212
  18 months (since last visit) | 0.778 (0.985)
  24 months (since last visit): number analyzed (Participants) | 188
  24 months (since last visit) | 0.553 (0.842)

4. Primary Outcome: Number of Visits in Outpatient Department by Study Visit
Description: Number of visits in outpatient department by study visit is reported. For the baseline visit mean and standard deviation of visits in outpatient department up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months mean and standard deviation of visits in outpatient department since the last study visit is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: visits per patient
Arm/Group | Idiopathic Pulmonary Fibrosis Diagnosed Patients
Number analyzed (Participants) | 301
visits per patient
  Baseline (up to 12 months prior to baseline visit) | 2.844 (3.042)
  3 months (since last visit): number analyzed (Participants) | 255
  3 months (since last visit) | 0.545 (0.899)
  6 months (since last visit): number analyzed (Participants) | 245
  6 months (since last visit) | 0.502 (0.852)
  12 months (since last visit): number analyzed (Participants) | 236
  12 months (since last visit) | 0.856 (1.358)
  18 months (since last visit): number analyzed (Participants) | 211
  18 months (since last visit) | 0.664 (1.217)
  24 months (since last visit): number analyzed (Participants) | 188
  24 months (since last visit) | 0.489 (0.939)

5. Primary Outcome: Number of Visits in Pulmonologists by Study Visit
Description: Number of visits in pulmonologists by study visit is reported. For the baseline visit mean and standard deviation of visits in pulmonologists up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months mean and standard deviation of visits in pulmonologists since the last study visit is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: visits per patient
Arm/Group | Idiopathic Pulmonary Fibrosis Diagnosed Patients
Number analyzed (Participants) | 301
visits per patient
  Baseline (up to 12 months prior to baseline visit) | 3.027 (2.209)
  3 months (since last visit): number analyzed (Participants) | 257
  3 months (since last visit) | 0.654 (0.839)
  6 months (since last visit): number analyzed (Participants) | 245
  6 months (since last visit) | 0.624 (0.777)
  12 months (since last visit): number analyzed (Participants) | 237
  12 months (since last visit) | 0.928 (1.171)
  18 months (since last visit): number analyzed (Participants) | 212
  18 months (since last visit) | 0.698 (1.05)
  24 months (since last visit): number analyzed (Participants) | 188
  24 months (since last visit) | 0.479 (0.749)

6. Primary Outcome: Number of Visits in Other Physicians Than the Pulmonologists by Study Visit
Description: Number of visits in other physicians than the pulmonologists by study visit is reported.
  For the baseline visit mean and standard deviation of visits in other physicians than the pulmonologists up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months mean and standard deviation of visits in other physicians than the pulmonologists since the last study visit is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: visits per patient
Arm/Group | Idiopathic Pulmonary Fibrosis Diagnosed Patients
Number analyzed (Participants) | 301
visits per patient
  Baseline (up to 12 months prior to baseline visit) | 1.056 (2.012)
  3 months (since last visit): number analyzed (Participants) | 253
  3 months (since last visit) | 0.34 (0.626)
  6 months (since last visit): number analyzed (Participants) | 243
  6 months (since last visit) | 0.358 (0.749)
  12 months (since last visit): number analyzed (Participants) | 237
  12 months (since last visit) | 0.561 (0.979)
  18 months (since last visit): number analyzed (Participants) | 211
  18 months (since last visit) | 0.588 (1.098)
  24 months (since last visit): number analyzed (Participants) | 188
  24 months (since last visit) | 0.505 (0.831)

7. Primary Outcome: Number of Idiopathic Pulmonary Fibrosis (IPF) Related Procedures by Study Visit
Description: Number of Idiopathic Pulmonary Fibrosis (IPF) related procedures by study visit is reported.
  For the baseline visit mean and standard deviation of Idiopathic Pulmonary Fibrosis (IPF) related procedures up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months mean and standard deviation of Idiopathic Pulmonary Fibrosis (IPF) related procedures since the last study visit is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IPF related procedures per patient
Groups:
- Idiopathic Pulmonary Fibrosis Patients: This arm includes all Idiopathic Pulmonary Fibrosis (IPF) diagnosed patients in Greece who participated in this study
Arm/Group | Idiopathic Pulmonary Fibrosis Patients
Number analyzed (Participants) | 301
IPF related procedures per patient
  Baseline (up to 12 months prior to baseline visit) | 2.638 (1.067)
  3 months (since last visit): number analyzed (Participants) | 259
  3 months (since last visit) | 1.216 (1.015)
  6 months (since last visit): number analyzed (Participants) | 247
  6 months (since last visit) | 1.271 (1.026)
  12 months (since last visit): number analyzed (Participants) | 237
  12 months (since last visit) | 1.722 (1.241)
  18 months (since last visit): number analyzed (Participants) | 212
  18 months (since last visit) | 1.613 (1.27)
  24 months (since last visit): number analyzed (Participants) | 188
  24 months (since last visit) | 1.569 (1.345)

8. Primary Outcome: Number of Patients in Each Category of Hospitalizations by Study Visit
Description: Number of patients in each category of hospitalizations by study visit is reported.
  For the baseline visit number of patients in each category of hospitalizations up to 12 months prior to baseline visit is reported.
  For the study visits at 3 months, at 6 months, at 12 months, at 18 months and at 24 months number of patients in each category of hospitalizations since the last study visit is reported.
  The categories of hospitalization were:
  * No
  * Yes
  * Unknown
  * Missing
Time Frame: At baseline up to 12 months prior to baseline visit) and at 3 months, at 6 months, at 12 months, at 18 months and at 24 months after the baseline visit.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Number analyzed (Participants) | 96 | 205
Participants
  Baseline (up to 12 months prior to baseline visit): No | 83 | 183
  Baseline (up to 12 months prior to baseline visit): Yes | 13 | 22
  Baseline (up to 12 months prior to baseline visit): Unknown | 0 | 0
  Baseline (up to 12 months prior to baseline visit): Missing | 0 | 0
  3 months (since last visit): No | 85 | 169
  3 months (since last visit): Yes | 1 | 5
  3 months (since last visit): Unknown | 0 | 1
  3 months (since last visit): Missing | 10 | 30
  6 months (since last visit): No | 80 | 162
  6 months (since last visit): Yes | 0 | 7
  6 months (since last visit): Unknown | 0 | 0
  6 months (since last visit): Missing | 16 | 36
  12 months (since last visit): No | 73 | 152
  12 months (since last visit): Yes | 3 | 9
  12 months (since last visit): Unknown | 0 | 0
  12 months (since last visit): Missing | 20 | 44
  18 months (since last visit): No | 72 | 132
  18 months (since last visit): Yes | 1 | 8
  18 months (since last visit): Unknown | 0 | 0
  18 months (since last visit): Missing | 23 | 65
  24 months (since last visit): No | 62 | 120
  24 months (since last visit): Yes | 2 | 5
  24 months (since last visit): Unknown | 0 | 0
  24 months (since last visit): Missing | 32 | 80

9. Primary Outcome: Number of Patients in Each Category With Usage of Pirfenidone and Nintedanib
Description: Number of patients in each category with usage of pirfenidone and nintedanib is reported.
  The categories for usage of pirfenidone and nintedanib are the following:
  * Yes
  * No
  * Unknown
  * Missing
Time Frame: From signing the informed consent onwards until the end of the study, up to 24 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Number analyzed (Participants) | 96 | 205
Participants
  Pirfenidone: Yes | 33 | 87
  Pirfenidone: No | 54 | 114
  Pirfenidone: Unknown | 0 | 0
  Pirfenidone: Missing | 9 | 4
  Nintedanib: Yes | 45 | 81
  Nintedanib: No | 41 | 116
  Nintedanib: Unknown | 0 | 0
  Nintedanib: Missing | 10 | 8

10. Secondary Outcome: Number of Patients in Each Category of Concomitant Medications
Description: Concomitant medication was defined as any treatment presented following the Informed Consent Form (ICF) signature. If stop date was missing in the electronic Case Report Form (eCRF), medication was considered as concomitant. The number of patients in each category of the following concomitant medications is reported. The concomitant medications are:
  * Corticosteroids
  * N-Acetylcysteine
  * Azathioprine
  * Cyclophosphamide
  * Cyclosporine A
  * Other immuno-suppressant
  * Anticoagulants
  * Gastroesophageal reflux disease (GERD) medication
  * Phosphodiesterase type 5 (PDE-5) inhibitor
  * Endothelin receptor antagonist
  * Non-steroidal anti-inflammatory drugs (NSAIDs) other than aspirin
  * Hormonal contraceptives
  * Hormone replacement therapy
  * Anti-vascular endothelial growth factor (VEGF) drugs
  * Other (other than listed above)
  The categories for each concomitant medication listed above are the following:
  * Yes
  * No
  * Unknown
  * Missing
Time Frame: From signing the informed consent onwards until the end of the study, up to 24 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
Number analyzed (Participants) | 96 | 205
Participants
  Corticosteroids: Yes | 11 | 21
  Corticosteroids: No | 73 | 175
  Corticosteroids: Unknown | 0 | 0
  Corticosteroids: Missing | 12 | 9
  N-Acetylcysteine: Yes | 1 | 3
  N-Acetylcysteine: No | 83 | 194
  N-Acetylcysteine: Unknown | 0 | 0
  N-Acetylcysteine: Missing | 12 | 8
  Azathioprine: Yes | 0 | 0
  Azathioprine: No | 84 | 197
  Azathioprine: Unknown | 0 | 0
  Azathioprine: Missing | 12 | 8
  Cyclophosphamide: Yes | 0 | 1
  Cyclophosphamide: No | 84 | 195
  Cyclophosphamide: Unknown | 0 | 0
  Cyclophosphamide: Missing | 12 | 9
  Cyclosporine A: Yes | 0 | 0
  Cyclosporine A: No | 84 | 195
  Cyclosporine A: Unknown | 0 | 0
  Cyclosporine A: Missing | 12 | 10
  Other immuno-suppressant: Yes | 0 | 4
  Other immuno-suppressant: No | 81 | 189
  Other immuno-suppressant: Unknown | 0 | 0
  Other immuno-suppressant: Missing | 15 | 12
  Anticoagulants: Yes | 34 | 67
  Anticoagulants: No | 53 | 129
  Anticoagulants: Unknown | 0 | 0
  Anticoagulants: Missing | 9 | 9
  GERD medication: Yes | 28 | 84
  GERD medication: No | 57 | 110
  GERD medication: Unknown | 0 | 0
  GERD medication: Missing | 11 | 11
  PDE-5 inhibitor: Yes | 0 | 5
  PDE-5 inhibitor: No | 83 | 189
  PDE-5 inhibitor: Unknown | 0 | 0
  PDE-5 inhibitor: Missing | 13 | 11
  Endothelin receptor antagonist: Yes | 0 | 2
  Endothelin receptor antagonist: No | 84 | 192
  Endothelin receptor antagonist: Unknown | 0 | 0
  Endothelin receptor antagonist: Missing | 12 | 11
  NSAIDs other than aspirin: Yes | 0 | 0
  NSAIDs other than aspirin: No | 84 | 194
  NSAIDs other than aspirin: Unknown | 0 | 0
  NSAIDs other than aspirin: Missing | 12 | 11
  Hormonal contraceptives: Yes | 0 | 0
  Hormonal contraceptives: No | 83 | 192
  Hormonal contraceptives: Unknown | 0 | 0
  Hormonal contraceptives: Missing | 13 | 13
  Hormone replacement therapy: Yes | 2 | 2
  Hormone replacement therapy: No | 81 | 188
  Hormone replacement therapy: Unknown | 0 | 0
  Hormone replacement therapy: Missing | 13 | 15
  Anti-VEGF drugs: Yes | 0 | 0
  Anti-VEGF drugs: No | 83 | 192
  Anti-VEGF drugs: Unknown | 0 | 0
  Anti-VEGF drugs: Missing | 13 | 13
  Other: Yes | 85 | 176
  Other: No | 0 | 0
  Other: Unknown | 0 | 0
  Other: Missing | 11 | 29

ADVERSE EVENTS:
Time Frame: From signing the informed consent onwards until the end of the study, up to 24 months.
Description: Full Analysis Set (FAS) comprised all subjects enrolled in the study with at least one measurement of any of the primary endpoints during the study. This population was used to run any statistics of the study.
Arm/Group | IPF Patients With Less Than 6 Months Diagnosis | IPF Patients With Equal or More Than 6 Months Diagnosis
All-Cause Mortality (participants affected / at risk) | 10/96 | 45/205
Serious Adverse Events (participants affected / at risk) | 7/96 | 22/205
Other Adverse Events (participants affected / at risk) | 10/96 | 21/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Patients With Less Than 6 Months Diagnosis (N=96) | IPF Patients With Equal or More Than 6 Months Diagnosis (N=205)
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 4
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 3
Septic shock (Infections and infestations) | 0 | 1
Transplantation complication (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Patients With Less Than 6 Months Diagnosis (N=96) | IPF Patients With Equal or More Than 6 Months Diagnosis (N=205)
Diarrhoea (Gastrointestinal disorders) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03074149/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03074149/SAP_001.pdf